CLINICAL TRIAL: NCT03237897
Title: Evaluation of a Preoperative Education Class for Colorectal Surgery Patients
Status: Withdrawn | Type: Observational
Why Stopped: Study withdrawn due to staff unavailability and limited resources
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 07-16-05E
Record Dates: First submitted 2016-09-23; First posted 2017-08-03 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Surgery
Keywords: ERAS; Enhanced recovery after surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Class attendees: A cohort of patients who are scheduled to undergo colorectal surgical procedures and attend the preoperative education class. Patients will be affixed with a pedometer in the postoperative period until discharge.
  Interventions: Behavioral: Preoperative education class; Behavioral: Pedometer
- Class non-attendees: A cohort of patients who are scheduled to undergo colorectal surgical procedures and do not attend the scheduled preoperative education class. Patients will be affixed with a pedometer in the postoperative period until discharge.
  Interventions: Behavioral: Pedometer

INTERVENTIONS:
Behavioral: Preoperative education class — The preoperative enhanced recovery after surgery education class will be offered twice a week in coordination with anesthesia preoperative appointments to minimize inconvenience for patients. Patients will need to attend only one class. All participants will be offered the class. This class will be one hour in duration and will be taught by a surgical advanced care practitioner familiar with the details of colorectal surgery. The class will include detailed information about preoperative care, intraoperative care, and postoperative care.
  Groups: Class attendees
Behavioral: Pedometer — A pedometer will be affixed to patients in the immediate postoperative period and removed at time of discharge

SUMMARY:
The purpose of the study is to evaluate the value and effectiveness of a newly-implemented preoperative education class for patients undergoing colorectal surgery.

DETAILED DESCRIPTION:
This is a non-randomized study to be conducted in a cohort of patients who are scheduled to undergo colorectal surgical procedures at Carolinas Medical Center (CMC)-Main. The primary objective of this study is to determine the effect of preoperative education classes on postoperative compliance with mobilization guidelines. Secondary objectives of this study are to evaluate the effect of the preoperative education class on patient knowledge, anxiety, and satisfaction, and postoperative outcomes such as inpatient length of stay, postoperative complications, and 30-day readmission rates. Data will be compared between patients who are scheduled to attend the class and attend and those who are scheduled to attend the class and do not.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo surgical operations of the colon or rectum at Carolinas Medical Center Main

Exclusion Criteria:

* A medical condition, laboratory finding, or physical exam finding that precludes participation
* Develop a significant intra- or postoperative complication that precludes or delays participation for longer than 4 weeks; or
* Have anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include only patients scheduled to undergo colorectal surgical procedures at CMC-Main.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Time to ambulation | from time of surgery until the time of first documented ambulation, assessed up to 90 days
  time to first ambulation following surgery measured by pedometer and notations made by nursing staff in the patient records prior to patient discharge.
Mean number of steps | from time of surgery until the time of discharge, up to 90 days
  mean number of steps taken daily as measured by pedometer

SECONDARY OUTCOMES:
Knowledge level | date of preoperative education class (up to 2 weeks prior to time of surgery) and date of first postoperative follow-up appointment (up to 90 days following surgery)
  Knowledge level assessed by knowledge survey administered to patients
Patient anxiety level | date of enrollment and date of discharge, up to 90 days following surgery
  Patient anxiety level assessed by anxiety survey administered to patients
Patient satisfaction score | date of first postoperative follow-up appointment, up to 90 days following surgery
  Patient satisfaction score assessed by satisfaction survey administered to patients
30-day readmission rate | 30 days following surgery
Inpatient length of stay | from date of surgery until the date of discharge, up to 90 days
  Inpatient length of stay measured in number of days

CONTACTS AND LOCATIONS:
Overall Officials: Caroline E Reinke, MD, Principal Investigator — Carolinas Medical Center

IPD SHARING:
Plan to Share IPD: Undecided